CLINICAL TRIAL: NCT03266029
Title: Single-Arm Observational Double - Blind Study Designed to Clinically Evaluate Cordio Application in Adult Patients With ADHF
Brief Title: Clinical Evaluation of Cordio App in Adult ADHF Patients
Status: Completed | Type: Observational
Sponsor: Cordio Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CA001
Record Dates: First submitted 2017-08-19; First posted 2017-08-29 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cordio App

SUMMARY:
Observational study on ADHF patients at one site in Israel. After signing informed consent and undergoing screening assessments, eligible patients will record sentences into a smartphone. The app will upload the vocal data to the sponsor's servers for analysis. The patient will record at hospital: admittion, release. Before hospital release, if applicable and upon patient agrreement, an app will be installed in a smartphone in order to continue the recording at home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHF (pulmonary congestion)
* Known diagnosis of HF, with either preserved or reduced LVEF.
* 18+ years old.
* Able to understand and provide written informed consent.

Exclusion Criteria:

* Subjects unable to comply with the daily use of the application due to mental disorders.
* GFR <25 ml/min who are non-responsive to diuretic therapy or who are on chronic renal dialysis.
* Subjects with congenital heart disease or mechanical right heart valve(s).
* Airway and lung infection and Sepsis
* Patients with severe alcohol or drug use.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitals/ CHF clinics
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2015-05-24 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
voice recording analysis - system is being developed to distinguish between 'dry' and 'wet' clinical state in ADHF patients (Speech Measure- SM- parameter) | 5 years
  Anyalysis of voice recordings; admission vs. discharge

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Azzam, Prof., Principal Investigator — Rambam Health Care Facility
Locations (1):
- Rambam Health Care Facility, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amir O, Abraham WT, Azzam ZS, Berger G, Anker SD, Pinney SP, Burkhoff D, Shallom ID, Lotan C, Edelman ER. Remote Speech Analysis in the Evaluation of Hospitalized Patients With Acute Decompensated Heart Failure. JACC Heart Fail. 2022 Jan;10(1):41-49. doi: 10.1016/j.jchf.2021.08.008. Epub 2021 Dec 8. PMID 34969496